CLINICAL TRIAL: NCT00978003
Title: Vasti Control of Patellofemoral Kinematics in Asymptomatic Volunteers
Brief Title: Vasti Control of Patellofemoral Kinematics in Asymptomatic Volunteer
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 090217; 09-CC-0217
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-04

CONDITIONS: Abnormalities; Patellofemoral Pain Syndrome
Keywords: Maltracking; Anterior Knee Pain; Knee; Natural History
MeSH Terms: conditions — Congenital Abnormalities; Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Healthy Volunteers: Adults age 18-55.

SUMMARY:
Background:

* Patellofemoral pain syndrome is one of the most common knee problems. It is characterized by pain in the front of the knee that is aggravated by deep knee flexion, prolonged sitting, and repetitive movement. The most widely accepted theory regarding the source of this pain is that a force imbalance around the knee puts extra stress on the area, leading to pain.
* Researchers are interested in learning more about the muscle groups around the knee to better understand the causes of knee pain.

Objectives:

- To obtain more information on how muscles, tendons, and bones work together to cause motion in the knee, both in the normal state and after immobilizing certain muscles around the knee.

Eligibility:

- Healthy individuals between the ages of 18 and 55, who have no current or chronic muscle, bone, or joint problems and who have no implants or other problems that would prevent them from receiving a magnetic resonance imaging (MRI) scan.

Design:

* This protocol will be carried out over two visits, both of which will involve using standard MRI sequences to look at the knee at rest and in motion.
* The first part will examine the knee under its natural state, with a standard MRI scan of the knee both at rest and in motion.
* The second part will involve temporarily reducing the force producing capabilities of one of the extensor muscles in the knee. To do so, study doctors will inject lidocaine into the muscle, which will temporarily (for approximately 2 hours) block the force producing capacity of this muscle, and then perform the MRI scan....

DETAILED DESCRIPTION:
Patellofemoral pain syndrome is one of the most common problems of the knee. It is characterized by anterior knee pain that is aggravated by deep knee flexion, prolonged sitting, and repetitive flexion/extension. The most widely accepted theory in regards to the source of this pain is that a force imbalance around the knee leads to static patellofemoral malalignment and dynamic patellofemoral maltracking. In turn, this malalignment and maltracking lead to elevated joint contact stresses, which ultimately leads to patellofemoral pain. Current understanding of patellofemroal maltracking is typically focused on static 2D alignment (lateral tilt and displacement). Yet, patellofemoreal pain is most often exacerbated during dynamic events and the patella has complete six degrees of freedom in its movement. More recent studies have been able to quantify patellofemoral kinematics during volitional dynamic tasks and demonstrate that the maltracking problem is more complex than originally postulated. Specifically, in patients with patellofemoral pain, altered kinematics are not limited to excessive patellar lateral translation and tilt, but include excessive patellar superior translation along with excessive flexion and varus rotation. Although these results are useful in demonstrating how specific maltracking patterns could lead to patellofemoral pain, they do not present any associations between a potentially altered force balance around the knee and the observed maltracking patterns. Therefore, the overall goal of this work is to determine the specific sources of maltracking patterns in patellofemoral pain. As part of this overall goal, the purpose of this study is to determine how the loss of force in the vasti medialis muscle alters the dynamic control of patellar kinematics.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Healthy male and female volunteers between the ages of 18 and 55.

<TAB>

EXCLUSION CRITERIA:

1. Any relevant medical problems (connective tissue problems, active arthritis, etc.)
2. Any clinical signs of a knee impairment in the joint being studied, including abnormal range of motion, muscle weakness, malaligment, and ligament damage.
3. Any serious injury to the joint being studied, previous surgery on the joint being studied or extreme pain at the joint being studied.
4. Allergy/hypersensitivity to lidocaine.
5. Liver disease.
6. Open angle glaucoma.
7. Cardiac arrhythmias, congenital heart disease.
8. G6PD.
9. Any female who is pregnant.

A volunteer will be excluded if they have a contraindication to MR imaging. Examples include:

1. Metal within their body, which might be expected to concentrate radiofrequency fields or cause tissue damage from twisting in a magnetic field (e.g., aneurysm clip, implanted neural stimulator, implanted cardiac pacemaker or autodefibrillator, cochlear implant, ccular foreign body (e.g. metal shavings, insulin pump).
2. A condition, which would preclude them from participating in an MR imaging study (e.g., paralyzed hemidiaphragm, morbid obesity, severe claustrophobia).
3. A condition that presents an unnecessary risk to them or their unborn child (e.g., pregnancy, previous surgery of uncertain type, symptoms of pheochromocytoma or insulinoma).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects for this study will be recruited through the Patient Recruitment and Public Liaison (PRPL) office. PRPL will respond to clinical research study inquiries, conduct preliminary screening for the protocol, and refer prospective patients to the Protocol Manager.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-10-22 (Actual)

PRIMARY OUTCOMES:
Eliminating the force producing capacity of the VM will increase patellar lateral shift, lateral tilt and valgus rotation. | End of study
  MRI imaging followed by muscle block and ultrasound.

SECONDARY OUTCOMES:
The amount of increase in patellar lateral shift, lateral tilt and valgus rotation, seen with the loss of the VM muscle will be correlated with the inferior- superior position of the patella relative to the femur. | End of study
  MRI imaging followed by muscle block and ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Frances T Gavelli, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-CC-0217.html